CLINICAL TRIAL: NCT04393441
Title: A Multicenter, Single-masked, Randomized Study to Compare the Efficacy and Safety of a New Artificial Tear Formulation (011516X) With Systane® Ultra Multidose for 90 Days in Participants With Dry Eye Disease
Brief Title: Efficacy and Safety of a New Artificial Tear Formulation Compared With Systane Ultra Multidose in Participants With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-301-005
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye Disease (DED)
Keywords: Dry Eye Disease; DED
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systane® Ultra Multidose (Active Comparator): All participants administered 1 to 2 drops of REFRESH PLUS® 3 times daily in each eye for approximately 7 days during a run-in period prior to randomization on Day 1. Participants then administered 1 to 2 drops of Systane® Ultra Multidose in each eye 3 times daily for up to 90 days.
  Interventions: Drug: Systane Ultra Multidose; Drug: REFRESH PLUS®
- 011516X (New Artificial Tear Formulation) (Experimental): All participants administered 1 to 2 drops of REFRESH PLUS® 3 times daily in each eye for approximately 7 days during a run-in period prior to randomization on Day 1. Participants then administered 1 to 2 drops of 011516X in each eye 3 times daily for up to 90 days.
  Interventions: Drug: 011516X (New Artificial Tear Formulation); Drug: REFRESH PLUS®

INTERVENTIONS:
Drug: 011516X (New Artificial Tear Formulation) — Topical eye drops
  Arms: 011516X (New Artificial Tear Formulation)
Drug: Systane Ultra Multidose — Topical eye drops
  Arms: Systane® Ultra Multidose
Drug: REFRESH PLUS® — Topical eye drops
  Other Names: 8197X

SUMMARY:
The purpose of this study is to compare the efficacy and safety of a new artificial tear formulation (011516X) with Systane® Ultra Multidose for 90 days in participants with Dry Eye Disease (DED).

ELIGIBILITY:
Inclusion Criteria:

* At the Screening (Day -7) and Baseline (Day 1) visits, at least 1 eye must qualify based on corneal and conjunctival staining scores
* Have used an artificial tear product for DED within 6 months of the Screening (Day -7) visit
* Have ability/agreement to continue to wear existing current spectacle correction during the study period (if applicable)
* If using any form of topical ophthalmic cyclosporine (i.e., RESTASIS®) or lifitegrast 5% ophthalmic solution (Xiidra®), participants must be using the drops for ≥90 days prior to the Screening (Day -7) visit and plan to continue without change for the duration of the study
* A female participant is eligible to participate if she is not pregnant (i.e., has a negative in-office urine pregnancy test at Screening [Day -7] and does not verbally report pregnancy at the Day 1 [Baseline] visit; is not breastfeeding, and at least 1 of the following conditions applies:

  1. A woman not of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance for the duration of the study

Exclusion Criteria:

* Have uncontrolled severe systemic disease that, in the assessment of the investigator, would put safety of the participant at risk through participation, or which would prevent or confound protocol-specified assessments (eg, hypertension and diabetes, Sjögren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, immunodeficiency disease, etc.)
* Participant has worn contact lenses in the last 90 days prior to the Screening (Day -7) visit and/or participant anticipates contact lens wear during the study
* Have any scheduled or planned systemic surgery or procedure during the study, which in the investigator's opinion, may impact the participant's study participation
* Presence of 1 or more of the following ocular conditions:

  * Active ocular infection or non-keratoconjunctivitis sicca (KCS) ocular inflammation
  * Active ocular allergy
  * History of recurrent herpes keratitis or active disease within 6 months prior to the Screening (Day -7) visit
  * Corneal disorder or abnormality that affects corneal sensitivity or normal spreading of the tear film (except superficial punctate keratitis)
  * Severe blepharitis or obvious inflammation of the lid margin, which in the judgment of the investigator, may interfere with the interpretation of the study results
  * Keratoconjunctivitis sicca secondary to the destruction of conjunctival goblet cells, such as occurs with vitamin A deficiency or scarring such as that with cicatricial pemphigoid, alkali burns, Stevens-Johnson syndrome, trachoma, or irradiation
  * Substantial non-KCS keratitis with overlying corneal stain or other significant corneal findings not directly related to DED; in addition, participants with DED signs/symptoms (eg, filamentary keratitis) of a severity where topical monotherapy with an artificial tear would be inappropriate
* The start date of any systemic medication (including over-the-counter [OTC], herbal, prescription, or nutritional supplements) which may affect Dry Eye Disease (DED) or vision is <90 days prior to the Screening (Day -7) visit or a change in dosage is anticipated during the study.

Systemic medications, which may affect DED or vision, include but are not limited to the following: flax seed oil, fish oil, omega-3 supplements, cyclosporine, antihistamines, cholinergic agents, anticholinergics, antimuscarinics, beta blocking agents, tricyclic antidepressants, phenothiazines, estrogen, progesterone, and other estrogen derivatives

* Have occlusion of the lacrimal puncta for either eye, with punctal plugs or cauterization < 6 months prior to the Screening (Day -7) visit or anticipated use of such procedures during the study
* Use of lid-heating therapy (i.e., LipiFlow®, iLUX®, etc.), Meibomian gland probing, or therapeutic Meibomian gland expression in either eye < 6 months prior to the Screening visit (Day -7) or anticipated use during the study
* Have history of ocular/ophthalmic surgery or trauma, which could affect corneal sensitivity and/or tear distribution (eg, cataract surgery, laser-assisted in situ keratomileusis [LASIK], photorefractive keratectomy, or any surgery involving a limbal or corneal incision) within 12 months prior to the Screening (Day -7) visit
* Are currently using topical ocular medication (OTC, herbal or prescription) or TrueTear® (intranasal neurostimulator), or have used topical ocular medication (OTC, herbal or prescription) or TrueTear within 1 month of the Screening (Day -7) visit or plan use of such treatments during the study. Exception: participants who are using the following can be considered:

  * Marketed artificial tear product for the management of DED, which must be discontinued at the Screening (Day -7) visit
  * Monotherapy for glaucoma or ocular hypertension (OHT) using a prostaglandin analog, beta blocker, alpha-2 agonist, or carbonic anhydrase inhibitor; any topical intraocular pressure (IOP)-lowering medications must have a start date of ≥ 90 days prior to the Screening (Day -7) visit and dosage is not expected to change during the study
  * Cyclosporine topical ophthalmic preparation (eg, RESTASIS or other ophthalmic form) or lifitegrast 5% ophthalmic solution (Xiidra), with a start date of ≥ 90 days prior to the Screening (Day -7) visit and dosage is not expected to change during the study NOTE: Participants currently being treated with BOTH an IOP-lowering medication and topical ocular cyclosporine or lifitegrast cannot be enrolled.
* Are currently enrolled in an investigational drug or device study or participation in such a study within 30 days of entry into this study at the Screening (Day -7) visit
* Report an average daily artificial tear use of >6 times per day within 6 months of the Screening (Day -7) visit
* Females who are pregnant, nursing, or planning a pregnancy during the study or females who are of childbearing potential and not using a reliable method of contraception
* Have history of allergies or sensitivity to the study interventions or its components (including all REFRESH and Systane product lines) or diagnostics (eg, topical ocular anesthetic, sodium fluorescein, or lissamine green).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Robinson, MD, Study Director — Allergan
Locations (26):
- United States (26):
  - Milton M. Hom, OD, FAAO, Azusa, California
  - Global Research Management, Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Eric M. White OD Inc, San Diego, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Nature Coast Clinical Research, Crystal River, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Georgia Eye Partners, Atlanta, Georgia
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Kannarr Eye Care, LLC, Pittsburg, Kansas
  - Senior Health Services, Louisville, Kentucky
  - Moyes Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, Saint Charles, Missouri
  - Eye Care Associates of Nevada, Sparks, Nevada
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Wake Forest Health Network Ophthalmology - Oak Hollow, High Point, North Carolina
  - Eye Care Associates of Greater Cincinnati, Inc. dba Apex Eye, Cincinnati, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, Nashville, Tennessee
  - DCT-Shah Research, LLC dba Discovery Clinical Trials, Mission, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Systane® Ultra Multidose | 011516X (New Artificial Tear Formulation)
Started | 200 | 200
Safety Population (Safety Population consisted of all treated participants who received/took ≥1 administration of study intervention.) | 199 | 200
Completed | 192 | 186
Not Completed | 8 | 14
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Deviation | 2 | 1
Not completed — Reason not Specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intend to treat (ITT) population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane® Ultra Multidose | 011516X (New Artificial Tear Formulation) | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.95) | 59.3 (13.55) | 58.4 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 157 | 323
  Male | 34 | 43 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 33 | 65
  Not Hispanic or Latino | 168 | 167 | 335
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 12 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 30 | 79
  White | 147 | 157 | 304
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Total Staining Score in the Study Eye [Mean (Full Range); unit: score on a scale] — Total staining score=sum of corneal and conjunctival staining score using Modified National Eye Institute/Industry Workshop(NEI) grading scale.Cornea is divided into 5 zones, nasal and temporal conjunctiva is divided into 6 zones.Combined total staining score=sum of five zones on cornea and six zones on conjunctiva. Each zone is graded on a 0 to 5 scale(0=no staining;1=trace;2=mild;3=moderate;4=severe;5=very severe), total score ranges=0 to 55.Higher score=worst dry eye condition. Study eye=worst eye based on total ocular staining score at Baseline.
  score on a scale | 13.4 [6 to 35] | 12.8 [6 to 37] | 13.1 [6 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Staining Score at Day 90 in the Study Eye
Description: The total staining score is the sum of corneal and conjunctival staining score using Modified NEI grading scale. The cornea is divided into 5 zones and the nasal and temporal conjunctiva is divided into 6 zones. The combined total staining score is based on the sum of the five zones on the cornea and six zones on the conjunctiva. Each zone is graded on a 0 to 5 scale (0=no staining; 1=trace; 2=mild; 3=moderate; 4=severe; 5=very severe), for a total score ranging from 0 to 55. The higher the score, the worse the dry eye condition. A negative change from Baseline represents a decrease in the severity of staining (improvement). The study eye is defined as the worst eye based on total ocular staining score at Baseline (Day 1). The fellow eye is the other eye. A mixed-effects model repeated measures (MMMR) was used for analyses.
Time Frame: Baseline (Day 1) and Day 90
Population: ITT population consisted of all randomized participants. Overall number analyzed are the number of participants with data available for analyses at the given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Systane® Ultra Multidose | 011516X (New Artificial Tear Formulation)
Number analyzed (Participants) | 192 | 186
Number analyzed (eyes) | 192 | 186
score on a scale | -4.5 (0.40) | -3.4 (0.41)
Statistical Analysis 1: Comparison: Systane® Ultra Multidose vs 011516X (New Artificial Tear Formulation); Change from Baseline in Total Staining Score at Day 90: The null hypothesis was that 011516X tear formulation was to be considered noninferior to Systane Ultra MD if the upper limit of 2-sided confidence interval (CI) was less than 2.3 units; Test type: Non-Inferiority — MMRM with fixed effects=treatment, visit, visit by treatment interaction,Baseline total staining stratum(TSS),and Baseline TSS by visit interaction; p = 0.0475, MMRM; Least Squares Mean Difference = 1.1, 95% CI 2-sided [0.01 to 2.27], Standard Error of Mean 0.57

2. Secondary Outcome: Change From Baseline in Current Symptom Survey Total Score at Day 90
Description: The Current Symptom Survey is a self-assessed 6-item visual analog scale (VAS) survey that assesses symptoms of dry eye disease (DED) including: burning, dryness, irritation, grittiness/foreign body sensation, blurry/fluctuating vision, overall ocular pain/discomfort. Each individual symptom is rated using a score range of 0=none to 100=maximum. The total score, ranging from 0 to 600, is calculated as the sum of individual symptom scores. A negative change from Baseline indicates improvement in DED symptoms experienced by the participant. This is an overall evaluation not per eye. A MMMR model was used for analyses.
Time Frame: Baseline (Day 1) and Day 90
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Systane® Ultra Multidose | 011516X (New Artificial Tear Formulation)
Number analyzed (Participants) | 192 | 186
score on a scale | -138.5 (11.46) | -136.5 (11.62)
Statistical Analysis 1: Comparison: Systane® Ultra Multidose vs 011516X (New Artificial Tear Formulation); Test type: Other — No formal hypothesis was planned. The p-value for treatment differences is reported for reference; p = 0.9001, MMRM; MMRM with fixed effects=treatment, visit, visit by treatment interaction, Baseline TSS, and Baseline TSS by visit interaction; Least Squares Mean Difference = 2.1, 95% CI 2-sided [-30.03 to 34.14], Standard Error of Mean 16.32

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days post last dose (up to approximately 147 days)
Description: All-cause Mortality: ITT population consisted of all randomized participants; Serious Adverse Events and Other Adverse Events: Safety Population consisted of all treated participants who received/took ≥1 administration of study intervention.
Arm/Group | Systane® Ultra Multidose | 011516X (New Artificial Tear Formulation)
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 1/199 | 0/200
Other Adverse Events (participants affected / at risk) | 0/199 | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Systane® Ultra Multidose (N=199) | 011516X (New Artificial Tear Formulation) (N=200)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04393441/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT04393441/SAP_001.pdf